CLINICAL TRIAL: NCT05960552
Title: Establishment and Verification of Clinical Thinking Flowchart of Rescue Transesophageal Echocardiography in the Diagnosis and Treatment of Perioperative Patients in Intensive and Critical Status
Brief Title: Perioperative Rescue Transesophageal Echocardiography in Intensive and Critical Status
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: K3052
Record Dates: First submitted 2023-07-06; First posted 2023-07-25 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Transesophageal Echocardiography
Keywords: Transesophageal Echocardiography; Surgery; Rescue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The PReTEE group (Experimental): Prior to clinical application of PReTEE, all participants designated must receive professional training. Within the given 120 seconds participants in the PreTEE group need to provide the leading cause with regard to difficult separation from cardiopulmonary bypass among high-risk cardiac surgical procedures.
  Interventions: Diagnostic Test: The PReTEE group
- The conventional TEE group (Active Comparator): The routine intra-operative TEE examinations are performed within the given 120 seconds before patients are separated from the cardiopulmonary bypass.
  Interventions: Diagnostic Test: The conventional TEE group

INTERVENTIONS:
Diagnostic Test: The PReTEE group — Prior to clinical application of PReTEE, all participants designated must receive professional training. They need to receive lectures focusing on the clinical thinking flowchart of rescue transesophageal echocardiography, in conjuntion with the simulator-based training. The discriminating ability of PReTEE will be further assessed in real clinical scenario, that is, within the specified 120 seconds participants in the PreTEE group need to provide the leading causes with regard to difficult separation from cardiopulmonary bypass in high-risk cardiac surgical procedures. All examinations will be supervised by a TEE expert owning to safety considerations but without help in views acquirement or interpretation. After completion of study assessments, the TEE expert will perform a standard comprehensive TEE, the results of which was reported to the attending cardiac anesthesiologist in charge of the patient and the recorders.
  Arms: The PReTEE group
Diagnostic Test: The conventional TEE group — Before cardiopulmonary bypass separation, conventional TEE examinations will be performed within the specified 120 seconds. Then, the expert will also perform a standard comprehensive TEE; the leading cause should also be presented to the attending anesthesiologists and recorders.
  Arms: The conventional TEE group

SUMMARY:
We initiate this study to assess the diagnostic efficiency of PReTEE, a simplified TEE scan sequence with a combination of 3 valuable views of ME 4C, ME AV LAX and TG SAX, in identifying cardiac pathologies in the phase of difficult cardiopulmonary bypass separation among patients who will undergo high-risk cardiac surgical procedures.

DETAILED DESCRIPTION:
There are 6 TEE operators who will participate in our trial, which is of restriction.

Also, the participants we scheme to include are all junior TEE operators at our institute, who have already skilled at images obtainment and interpretation. Prior to the trial initiation, all these TEE operators will be randomly assigned into either the PReTEE group or the conventional TEE group with a 1:1 ratio (3 per group). Due to another limitation of eligible patients, TEE examinations thereby for patients are not conducted by equal numbers of operators stratified by groups. Furthermore, patients will be examined by 1-4 operators and 1 expert without removing the probe when separated from cardiopulmonary bypass. The ultimate sample size we calculate is 46 TEE examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 yr and greater;
2. High-risk cardiac surgery (one of the followings): Baseline left ventricular ejection fraction < 50%, Coronary artery bypass graft combined with valve procedures, Multiple valve procedures (≥ 2), Aortic root or arch involved, Euroscore > 6, Previous cardiovascular surgery

Exclusion Criteria:

1. Lack of patient consent;
2. Esophageal pathology (stricture, tumor, perforation/laceration, ulcer or fistula, diverticulum);
3. Hiatus hernia; Perforated viscus;
4. Active/recent upper gastrointestinal (GI) bleed;
5. Non-elective cardiac procedures;
6. Preoperative mechanical cardiac support (ECMO, LVAD or IABP)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time taken in seconds in seeking out the leading cause of difficult CPB separation. | From the time of appearance of midesophageal 4 chamber view until the time of discrimination of the leading cause of difficult separation from cardiopulmonary bypass by the TEE operator, assessed up to 120 seconds.
  Time will be recorded in rea-time fashion from the appearance of midesophageal 4 chamber view to the diagnose of leading cause of difficult CPB separation in both the PReTEE group and the conventional group.
The rate of successful diagnosis. | From the time of appearance of midesophageal 4 chamber view until the time of discrimination of the leading cause of difficult separation from cardiopulmonary bypass by the TEE operator, assessed up to 120 seconds.
  Following the completion of TEE assessment by operators in the PreTEE group or in the conventional TEE group, the TEE expert in our center will then perform a standard comprehensive examination. The TEE expert will also be required to provide the leading cause of difficult separation, which then be presented to the attending anesthesiologist and cardiac surgeons as the reference of therapeutic approaches. The successful diagnosis is defined as the agreement of cause between operators in the PreTEE group or in the conventional TEE group and the expert.

SECONDARY OUTCOMES:
Detection rate of hypovolemia | From the time of appearance of midesophageal 4 chamber view until the time of discrimination of the leading cause of difficult separation from cardiopulmonary bypass by the TEE operator, assessed up to 120 seconds.
  Reduction in the LV cavity indicates hypovolemia.
Detection rate of left ventricular outflow tract obstruction | From the time of appearance of midesophageal 4 chamber view until the time of discrimination of the leading cause of difficult separation from cardiopulmonary bypass by the TEE operator, assessed up to 120 seconds.
  The occurrence of SAM
Detection rate of regional wall motion abnormality | From the time of appearance of midesophageal 4 chamber view until the time of discrimination of the leading cause of difficult separation from cardiopulmonary bypass by the TEE operator, assessed up to 120 seconds.
  Regional wall motion is commonly classified as 1) normal or hyperkinetic, 2) hypokinetic (reduced thickening), 3) akinetic (absence of thickening), and 4) dyskinetic (systolic thinning or aneurysmal changes
Detection rate of left ventricular systolic dysfunction | From the time of appearance of midesophageal 4 chamber view until the time of discrimination of the leading cause of difficult separation from cardiopulmonary bypass by the TEE operator, assessed up to 120 seconds.
  Left ventricular systolic dysfunction can be assessed as a reduction in systolic function and an increase in diastolic dimension.
Detection rate of right ventricular systolic dysfunction | From the time of appearance of midesophageal 4 chamber view until the time of discrimination of the leading cause of difficult separation from cardiopulmonary bypass by the TEE operator, assessed up to 120 seconds.
  A TEE with a D-shaped LV on trans-gastric short axis view is suggestive of RV volume overload and systolic dysfunction
Detection rate of right ventricular outflow tract obstruction | From the time of appearance of midesophageal 4 chamber view until the time of discrimination of the leading cause of difficult separation from cardiopulmonary bypass by the TEE operator, assessed up to 120 seconds.
  The occurrence of pulmonary embolism, residual thrombus or tumor is seen in the RA/ RV, leftward shift of the interatrial septum or moderate to severe tricuspid regurgitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Wang C, Tian Y, Bai B, He K, Lu H, Yu C, Miao Q. Application of a simplified transesophageal echocardiography examination sequence in high-risk cardiac surgery. Trials. 2024 Aug 13;25(1):535. doi: 10.1186/s13063-024-08338-9. PMID 39138581